CLINICAL TRIAL: NCT06647368
Title: Investigating the Effect of Glucagon on Cognitive Function and Cerebral Glucose Metabolism in Humans: A Pilot study_A
Brief Title: Development of a Non-invasive Method for Quantifying Cerebral Glucose Metabolism for Studying the Effect of Glucagon in Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolai Jacob Wewer Albrechtsen (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Sponsor-Investigator, Nicolai Jacob Wewer Albrechtsen, Principal Investigator, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GluCoMet_pilotA
Record Dates: First submitted 2024-10-14; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Glucose Metabolism
MeSH Terms: interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET with 18-FDG (Experimental)
  Interventions: Other: PET with 18-FDG

INTERVENTIONS:
Other: PET with 18-FDG — The intervention is a 1,5 hour PET scan, which will be performed in three steps (heart scan, brain scan and heart scan) and administration of radioactively labelled glucose (18-FDG) in two doses.

SUMMARY:
The aim of the study is to develop a non-invasive method for quantifying cerebral glucose metabolism by PET scans in humans. This method will be used in subsequent studies, where the effect of the pancreatic hormone glucagon on cerebral glucose metabolism will be studied.

The golden standard for quantifying cerebral glucose metabolism by PET scans is based on arterial blood sampling, which complicates research setup. This study will investigate if image derived measurements instead of arterial blood samples can be used to quantify cerebral glucose metabolism.

We will compare the calculations of cerebral glucose metabolism based on arterial blood samples and image derived measurements and hopefully these will correlate.

Healthy participants will be included, and each participant will participate in one study day, which includes intravenous administration of radioactively labelled glucose (18-FDG), arterial blood sampling and PET scans.

DETAILED DESCRIPTION:
Participants will arrive after a four hour fast. An arterial cannulation will be placed in the radial or brachial artery for blood sampling. A venous catheter will be placed in the antecubital vein for administration of 18-FDG. Blood glucose is measured.

Before administration of 18-FDG a "low dose" CT scan of the heart and brain will be performed.

At time 0 minutes 20 MBq 18-FDG will be administered, 10 minutes automatic blood sampling (from the arterial cannulation) will be started and a 10 minutes three part dynamic PET scan of the heart will be performed.

Approximately at time 20 minutes 180 MBq 18-FDG will be administered and a 40 minutes three part dynamic PET scan of the brain will be performed. During the first 10 minutes of the brain scan automatic blood sampling (from the arterial cannulation) will be performed and thereafter manual blood sampling will be performed every 5 minutes.

After the 40 minutes brain PET scan a 5 min post scan of the heart will be performed.

Radioactivity will be measured in the arterial blood samples and the results will be used for an Arterial Input Function (AIF).

Radioactivity measurements derived from the heart scans will be used for an Image Derived Input Function (IDIF).

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the participant information and signing the consent form
* Between 25 and 70 years of age
* Body mass index <= 25 kg/m^2

Exclusion Criteria:

* Enrolment in other research project that might interfere with the study
* Diabetes diagnosis
* Pregnancy or breastfeeding
* Use of medications which, in the opinion of the investigator, may jeopardise participant's safety or compliance with the protocol
* Diagnosis of psychiatric disorders, dementias, or any other neurological disorders that in the opinion of the investigator precludes compliance with the study protocol, evaluation of the results or represents an unacceptable risk for the participants safety
* Severe claustrophobia
* Cardiac problems including any of the following:

  1. Classified as being in New York Heart Association (NYHA) class III or IV
  2. Angina pectoris (chest pain) within the last 6 months
  3. Acute myocardial infarction (heart attack) within last 2 years
* Inadequately treated blood pressure at screening defined as repeated resting blood pressure outside the range 90-150 mmHg for systolic and 50-100 mmHg for diastolic.
* Active or recent malignant disease
* Current or history of severe alcohol use or drug/chemical abuse as per investigator's judgement
* Any chronic disorders or severe diseases which, in the opinion of the investigator, might jeopardise participant's safety or compliance with the protocol

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-10-22 (Estimated); Primary Completion 2024-12-17 (Estimated); Study Completion 2024-12-17 (Estimated)

PRIMARY OUTCOMES:
Tmax correlation | From administration of 180MBq 18-FDG and during the approximately first 15 min of the brain PET scan
  Difference between the blood-brain glucose transfer capacity (Tmax) calculated based on the image derived input function and Tmax calculated based on the arterial input funcion.

SECONDARY OUTCOMES:
CMRglc correlation | From administration of 180MBq 18-FDG and during the 40 min brain PET scan
  Difference between cerebral metabolic rate of glucose (CMRglc) calculated based on the image derived input function and CMRglc calculated based on the arterial input funcion.

CONTACTS AND LOCATIONS:
Overall Officials: Lisbeth Marner, MD PhD, Study Chair — University Hospital Bispebjerg and Frederiksberg; Nicolai J Wewer Albrecthsen, MD PhD, Principal Investigator — Department of Clinical Biochemistry, Copenhagen University Hospital - Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark
Locations (1):
- Department of Physiology and Nuclear Medicine, University of Copenhagen - Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark, Copenhagen, Denmark